CLINICAL TRIAL: NCT06122207
Title: A Randomized, Double-blind, Placebo-controlled Study to Confirm the Positive Effect of Fertibiome® (Ligilactobacillus Salivarius PS11610) on the Female Genital Tract Microbiota of Couples or Women With Fertility Disorders.
Brief Title: Effect of a Probiotic on the Female Genital Tract Microbiota of Participants With Fertility Disorders.
Acronym: PROFEC II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FEC/23.03
Record Dates: First submitted 2023-10-27; First posted 2023-11-08 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Fertility Disorders
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Women will take two daily doses containing approximately 2*10E9 Colony Forming Unit (CFU) of Ligilactobacillus salivarius PS11610 (Fertibiome®). Men will take one daily dose containing approximately 1*10E9 CFU of Ligilactobacillus salivarius PS11610 (Fertibiome®).
  In case of pregnancy during intervention, only women will continue taking 1 daily dose for the first 12 weeks of gestation.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Women will take two daily doses of Placebo supplement. Men will take one daily dose of Placebo supplement.
  In case of pregnancy during intervention, only women will continue taking 1 daily dose for the first 12 weeks of gestation.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — * Women: 1 capsule of probiotic (Ligilactobacillus salivarius PS11610) every 12 hours for 6-months. In case of pregnancy:
    * Women: 1 capsule of probiotic per day for 12 weeks.
  * Men: 1 capsule of probiotic (Ligilactobacillus salivarius PS11610) per day for 6-months.
  Arms: Probiotic
Dietary Supplement: Placebo — * Women: 1 capsule of placebo every 12 hours for 6-months. In case of pregnancy:
    * Women:1 capsule of placebo per day for 12 weeks.
  * Men: 1 capsule of placebo per day for 6-months.
  Arms: Placebo

SUMMARY:
In the last decades, numerous publications have broken the old paradigm that considered the urogenital tracts as sterile, demonstrating that microorganisms present in the urogenital tract represent the 9% of the whole human microbiome. Healthy urogenital microbiome improves implantation rate and pregnancy outcomes, whereas 40% of dysbiosis prevalence is observed in women under assisted reproductive treatment (ART).

Infertility causes are associated with male, female, or combined failure. It has been shown that oral probiotic treatment, mainly with Lactobacillus, recovers a healthy vaginal microbiota without safety concerns.

An interventional, randomized, double-blind, placebo-controlled study will be conducted to confirm the positive effect of the commercial probiotic product Fertibiome® on the vaginal dysbiosis of couples or women with fertility disorders.

The duration of the study will be of 6 months approximately, including 6 months of product intake. In case of pregnancy during intervention, women will continue their participation until week 12 of gestation.

Participants will be randomly assigned to one of the two study groups: control group with placebo administration or probiotic administration group. Women will take 1 capsule every 12 hours and men 1 per day. In case of women participating alone they will take 1 capsule every 12 hours. In case of pregnancy, only women will continue taking 1 capsule per day for the first 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Couples or women with ages between 18 and 40 for woman and between 18 and 55 for man (in case of couple participation).
* Couples or women with fertility disorders.
* Couples or women undergoing IVF treatment or willing to start it.
* Signature of the Informed Consent.

Exclusion Criteria:

* Women, not participating in the study with a couple, who have not undergone at least 4 cycles of artificial insemination with donor's sperm (AID) or 1 cycle of IVF without achieving evolutionary pregnancy.
* Women with Body Mass Index (BMI) ≥ 30.
* Couples where the woman has not infertility diagnosis while the man has any of the following characteristics:

  * Azoospermia
  * Sperm motility (A + B) < 25%.
  * Sperm morphology ≤ 2%.
  * Vas deferens obstruction.
* Couples or women with any of the following characteristics:

  * Chronic diseases that cause intestinal malabsortion.
  * Congenital or acquired immunodeficiency.
  * Current history or diagnosis of alcohol, tobacco, or drug abuse.
  * Uncertainty about the willingness or ability of participants to comply with the requirements of the protocol.
  * Under treatment with probiotics during the last week.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of women with vaginal dysbiosis after 3 months of treatment. | After 3 months of intervention.
  The percentage of vaginal dysbiosis confirmed will be compared between groups of treatment.
Percentage (%) of women with vaginal dysbiosis after 6 months of treatment. | After 6 months of intervention.
  The percentage of vaginal dysbiosis confirmed will be compared between groups of treatment.

SECONDARY OUTCOMES:
Number of vaginal dysbiosis criteria in case of pregnancy confirmation. | Up to 6 months.
Percentage (%) of women with vaginal dysbiosis. | Before intervention.
Number of dysbiosis criteria per woman. | Before intervention.
Number of dysbiosis criteria per woman. | After 3 months of treatment pregnancy confirmation.
Number of dysbiosis criteria per woman. | After 6 months of treatment or pregnancy confirmation.
Percentage of Lactobacillus in vaginal microbiota. | Before intervention.
Percentage of Lactobacillus in vaginal microbiota. | After 3 months of treatment or pregnancy confirmation.
Percentage of Lactobacillus in vaginal microbiota. | After 6 months of treatment or pregnancy confirmation.
Number of reproductive treatments during the study period. | After 6 months of treatment or pregnancy confirmation.
Pregnancy rate. | After 6 months of treatment or pregnancy confirmation.
Time elapsed from the beginning of the study, until the occurrence of pregnancy. | Up to 6 months.
Spontaneous pregnancy rate, not associated to fertility treatment (IVF or AI). | Up to 6 months.
Miscarriage rate in the first trimester of pregnancy. | Before 12 weeks of pregnancy.
Number of oocytes extracted. | Before IVF cycle.
Embryo Quality (A, B or C). | Before IVF cycle.
Number of vaginal dysbiosis criteria at the time of embryo transfer per IVF cycle. | Before IVF cycle.
Levels (pg/ml) of pro-inflammatory and anti-inflammatory markers in blood plasma of women. | Before intervention.
Levels (pg/ml) of pro-inflammatory and anti-inflammatory markers in blood plasma of women. | After 6 months of treatment or pregnancy confirmation.

CONTACTS AND LOCATIONS:
Locations (2):
- Dr. Miguel Raimundo (Portugal), Lisbon, Portugal
- Hospital Universitario La Paz, Madrid, Madrid, Spain